CLINICAL TRIAL: NCT06843148
Title: Stimulating Adipose Tissue Fatty Acid Disposal With Low-dose, Postprandial, Intermittent Niacin for the Treatment of Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD).
Brief Title: Stimulating Fat Tissue Storage With Niacin to Reduce Fat Accumulation in the Liver.
Acronym: AGL13
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre hospitalier universitaire de Québec- Université Laval (Unknown); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenure professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025-5648
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD); Liver Fibrosis/NASH; Non-Alcoholic Steato-Hepatitis (NASH)
Keywords: Fatty liver; Niacin; vitamin B3; nicotinic acid
MeSH Terms: conditions — Fatty Liver | interventions — Niacin; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): It will be a 12-week treatment phase. The placebo treatment will be administered once daily, at the end of the largest meal.
  Interventions: Drug: Placebo Oral Tablet
- Niacin group (Active Comparator): It will be a 12-week treatment phase. The treatment will be administered once daily, at the end of the largest meal.
  Interventions: Drug: Niacin (250mg)

INTERVENTIONS:
Drug: Niacin (250mg) — Niacin will be orally taken once daily with the largest meal. There will be a 3-week escalation period from 250 mg to 750 mg:
  * Week 1: 250mg
  * Week 2: 500mg
  * Week 3 to Week 12: 750mg (3 x 250mg caplets)
  Other Names: Nicotinic Acid; Vitamin B3
  Arms: Niacin group
Drug: Placebo Oral Tablet — Placebo will be orally taken once daily with the largest meal. There will be a 3-week escalation period from 250 mg to 750 mg:
  * Week 1: 250mg
  * Week 2: 500mg
  * Week 3 to Week 12: 750mg (3 x 250mg caplets)
  Arms: Placebo group

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) (aka non-alcoholic fatty liver disease), commonly occurring in individuals with obesity and type 2 diabetes can lead to liver inflammation/ fibrosis. MASLD results from fat being disproportionately deposited in the liver.

The goal of this mechanistic study is to investigate metabolic response in patients aged 50 to 80 years with non-alcoholic fatty liver disease, after niacin (vitamin B3) treatment.

The main questions it aims to answer are:

* Does Niacin lower the fat deposition in the liver?
* Does Niacin raise White Adipose Tissue storage of dietary fatty acids?

Researchers will compare Niacin to a placebo (a look-alike substance that contains no drug) to compare the metabolic response.

Duration of study per participant: Up to 28 weeks

DETAILED DESCRIPTION:
It will be a randomized crossover study with two 12-week treatment phases (niacin vs. placebo) with a 4-week washout period between the two treatment phases.

The two 12-week treatment phases will be performed in random order. The treatment will be administered once daily, at the end of the largest meal. There will be a 3-week dose escalation: from 250mg (the first week) to 750mg from week 3 onward.

The outcomes will be assessed at the end of each of these two treatment phases in all participants with metabolic visit A and B (i.e., a total of 4 metabolic visits).

Each metabolic visit will last 9 hours: it will be a test meal with perfusion of stable tracers, blood sampling, PET acquisitions using radiopharmaceuticals (18FTHA and 11C-palmitate) and MRI acquisitions.

The two visits A and B will be performed without and with acute administration of niacin with the test meal, respectively, to determine acute niacin-induced reduction in hepatic fatty acid flux.

The two visits will be performed at four to seven-day interval, in random order during the last week of each of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 80 years;
* diagnosed with MASLD, defined as the presence of liver steatosis + abdominal obesity (as defined by the International Diabetes Federation country/ethnic group-specific criteria;
* all women will be post-menopausal.

Exclusion Criteria:

1. Presence of advanced fibrosis (i.e., ≥ F3 based on liver stiffness > 10kPa) using vibration-controlled transient elastography (FibroScan), serum ALT > 3 times the normal upper limit, or signs of portal hypertension [106-109].
2. Other hepatic disease.
3. Previous diagnosis of diabetes.
4. Overt cardiovascular or renal disease, cancer (other than non-melanoma skin cancer), or other uncontrolled medical conditions.
5. Any contraindication to MRI.
6. Previous intolerance or allergy to nicotinic acid.
7. Having participated to a research study with exposure to radiation in the last two years before the start of the study.
8. Being allergic to eggs
9. Smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Prolonged small-dose niacin treatment does not lead to desensitization of the niacin-induced reduction in hepatic total fatty acids flux. | Week 12, Week 28
  Total 6 h integrated uptake of circulating NEFAs, DFAs, and all FAs in liver: represents the sum of the rate of NEFA uptake integrated over 360 min for the entire organ and the rate of DFA uptake integrated over 360 min for the entire organ.

SECONDARY OUTCOMES:
Change in White Adipose Tissue (WAT) and lean tissue Dietary Fatty Acid (DFA) uptake | Week 12, Week 28
  Determined from the same static (whole-body) acquisition image using oral administration of [18F]-Fluoro-6-Thia-Heptadecanoic Acid (FTHA)
Change in total hepatic fatty acid flux | Week 12, Week 28
  represents the sum of the rate of NEFA uptake and DFA uptake (PET scan using [18F]-FTHA and [11C]-palmitate
Change in hepatic Non-Esterified-Fatty-Acid (NEFA) uptake oxidation, esterification and secretion into very low-density lipoprotein (VLDL) | Week 12, Week 28
  [11C]-Palmitate PET. Calculated from the same multicompartmental equation using liver [11C]-palmitate kinetics
Change in Endogenous Glucose production and meal glucose systemic flux | Week 12, Week 28
  i.v. and oral stable isotope tracer
Change in plasma NEFA flux | Week 12, Week 28
  calculated from i.v. stable isotope tracer (mass spectrometry).
Change in hepatic Triglyceride (TG) content | Week 12, Week 28
  magnetic resonance imaging (MRI)
Change in insulin secretion | Week 12, Week 28
  Determined by measuring C-peptide kinetics following the liquid meal
Change in hormonal response | Week 12, Week 28
  Multiplex assay
Change in metabolite response | Week 12, Week 28
  Colorimetric assay
Change in plasma distribution of DFA metabolites | Week 12, Week 28
  calculated from i.v. and oral stable isotope tracers (mass spectrometry) incorporated into triglyceride-rich lipoproteins and NEFA.
Change in glycerol turnover | Week 12, Week 28
  calculated from [1,1,2,3,3-2H]-glycerol i.v.
Change in total substrate utilisation | Week 12, Week 28
  measured by using indirect calorimetry
Change in insulin resistance /sensitivity | Week 12, Week 28
  Determined by measuring circulating glucose, NEFA and insulin following the liquid meal.
Circulating markers of hepatic inflammation | Week1, Week 12, Week 16, Week 28
  Measurement of Alanine aminotransferase (ALT), Aspartate transaminase (AST) and platelet count for calculation of fibrosis-4 which is an index for liver fibrosis.
Adverse events | up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada